CLINICAL TRIAL: NCT03704051
Title: Breast Versus Bottle Study
Status: Completed | Type: Observational
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Alison Ventura, Associate Professor, California Polytechnic State University-San Luis Obispo
Other Study IDs: 2018-143-CO; R03HD096164 (NIH)
Record Dates: First submitted 2018-10-08; First posted 2018-10-12 (Actual); Results first posted 2022-11-15 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Breastfeeding; Bottle Feeding
Keywords: infant feeding; feeding interactions; maternal feeding practices; breastfeeding; bottle-feeding
MeSH Terms: conditions — Breast Feeding; Bottle Feeding

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breastfeeding First, then Bottle-feeding: Mother-infant dyads were observed while breastfeeding during their first visit to our laboratory and were observed while bottle-feeding expressed breast milk during their second visit to our laboratory.
  Interventions: Behavioral: Mode of Feeding (breastfeeding versus bottle-feeding)
- Bottle-feeding First, then Breastfeeding: Mother-infant dyads were observed while bottle-feeding expressed breast milk during their first visit to our laboratory and were observed while breastfeeding during their second visit to our laboratory.
  Interventions: Behavioral: Mode of Feeding (breastfeeding versus bottle-feeding)

INTERVENTIONS:
Behavioral: Mode of Feeding (breastfeeding versus bottle-feeding) — Infants will be breastfed during one lab visit and bottle-fed (with expressed breast-milk) during the other.

SUMMARY:
The objective of the proposed research is to conduct a within-subject experimental study that will assess the effect of feeding mode (breast- versus bottle-feeding) on the quality and outcome of infant feeding interactions.

ELIGIBILITY:
Inclusion Criteria:

* Mothers 18-40 years of age
* Infants 0-24 weeks of age
* Infants who have not yet been introduced to complementary foods and beverages
* Dyads are breast- and bottle-feeding
* Mother is predominantly or solely responsible for infant feeding

Exclusion Criteria:

* preterm birth (i.e., gestational age <37 weeks)
* low birth weight (<2500 g)
* maternal smoking during pregnancy
* current or past medical conditions that interfere with oral feeding
* history of slow growth or failure to thrive
* weight for length percentile <5th
* diagnosed developmental delay (e.g., Down's syndrome)

Ages: 0 Weeks to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A convenience sample of mother-infant dyads residing within 50 miles of California Polytechnic State University.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison K Ventura, PhD, Principal Investigator — Cal Poly
Locations (1):
- Healthy Kids Laboratory within the French Hospital Copeland Health Education Pavilion, San Luis Obispo, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not currently plan to make individual participant data available to other researchers.

REFERENCES:
- [Result] Ventura A, Hupp M, Lavond J. Mother-infant interactions and infant intake during breastfeeding versus bottle-feeding expressed breast milk. Matern Child Nutr. 2021 Oct;17(4):e13185. doi: 10.1111/mcn.13185. Epub 2021 May 3. PMID 33939269

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mothers of infants under 6 months of age were recruited through advertisements on social media platforms (e.g. Facebook and Instagram); advertisements in local Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) clinics; announcements in birthing, breastfeeding and parenting classes; and flyers displayed at local businesses.
Pre-assignment Details: There were no significant events in the study (for example, wash out, run-in) that occurred after participant enrollment, but prior to the first within-subject condition.
Groups:
- Breastfeeding First, Then Bottle-feeding: Mother-infant dyads in this group breastfed during the first visit, then bottle-fed expressed breast milk during the second visit.
- Bottle-Feeding First, Then Breastfeeding: Mother-infant dyads in this group bottle-fed expressed breast milk during the first visit, then breast-fed during the second visit.
Period: Overall Study
Arm/Group | Breastfeeding First, Then Bottle-feeding | Bottle-Feeding First, Then Breastfeeding
Started | 48 (24 mother-infant dyads (24 mothers + 24 infants = 48 participants total) participated in the first visit) | 46 (23 mother-infant dyads (23 mothers + 23 infants = 48 participants total) participated in the first visit)
Completed | 44 (2 mother-infant dyads (2 mothers + 2 infants = 4 participants total) in this group dropped out of the study after the first visit) | 46 (0 mother-infant dyads in this group dropped out of the study after the first visit)
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included mothers (n = 47) and their healthy infants <6 months of age (n = 47).
Groups:
- All Study Participants: This was a within-subject study; all mother-infant dyads (47 mothers + 47 infants = 94 participants total) were exposed to both conditions and the order of presentation was counterbalanced across dyads. Because all dyads were randomized to receive all interventions, all will be combined into one arm/group for the summary that follows.
  Mode of Feeding (breastfeeding versus bottle-feeding): Infants will be breastfed during one lab visit and bottle-fed (with expressed breast milk) during the other.
Arm/Group | All Study Participants
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: years] — Mother Age at Study Entry Population: Data are for mothers only (n = 47)
  years
    number analyzed (Participants) | 47
    (all) | 32.4 (4.2)
Age, Continuous [Mean (Standard Deviation); unit: months] — Infant Age at Study Entry Population: Data are for infants only (n = 47)
  months
    number analyzed (Participants) | 47
    (all) | 3.2 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data are for mothers only (n = 47)
  Participants
    number analyzed (Participants) | 47
    Female | 47
    Male | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data are for infants only (n = 47)
  Participants
    number analyzed (Participants) | 47
    Female | 20
    Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 70
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 86
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — All data collection took place in San Luis Obispo and Santa Barbara Counties, California
  participants
    United States | 94

OUTCOME MEASURES:

1. Primary Outcome: Infant Intake During the Observed Feeding (mL)
Description: For both breast- and bottle-feedings, infant intake will be assessed by pre- and post-weighing the baby on an infant scale (model 374; Seca, Hamburg, Germany). During bottle-feedings, we will also note whether the infant finishes the bottle.
Time Frame: 2-hour period
Measure: Mean (Standard Error); unit: mL
Units Other Than Participants: dyads
Groups:
- Breast- Versus Bottle-feeding: This was a within-subject study; all mother-infant dyads were exposed to both conditions: breastfeeding versus bottle-feeding with expressed breast milk
  Order of presentation was counterbalanced.
Arm/Group | Breast- Versus Bottle-feeding
Number analyzed (Participants) | 94
Number analyzed (dyads) | 47
mL
  Breastfeeding Condition | 91.9 (5.0)
  Bottle-feeding Condition | 87.6 (5.2)
Statistical Analysis 1: Comparison: Breast- Versus Bottle-feeding; Test type: Equivalence — A priori power analysis based on pilot testing with 12 dyads indicated that a sample size of at least 40 dyads would provide 80% power to detect significant within-subjects (condition, i.e., breastfeeding directly from the breast vs. bottle-feeding expressed breast milk) effects at an α = 0.05 Type I error level; p = 0.634, Mixed Models Analysis; All models adjusted for order of conditions, time since last feeding and infant age

2. Primary Outcome: Maternal Sensitivity to Infant Cues
Description: Mother and infant behavior during each feeding will be coded using the Nursing Child Assessment Parent-Child Interaction - Feeding Scale (NCAFS). This scale contains six subscales, four of which describe maternal attributes (Sensitivity to Cues, Response to Child's Distress, Social-Emotional Growth Fostering, and Cognitive Growth Fostering) and two of which describe infant attributes (Clarity of Cues and Responsiveness to Caregiver). The proposed analysis will focus on the Sensitivity to Cues subscale, which measures the degree to which the mother is able to understand and respond to her child's cues. This scale provides a global measure of how sensitive the mother is to the infant's needs during the feeding interaction. Possible score range is 0-16, which is derived from summing together maternal scores for each of the 16 subscale items. Higher scores indicate greater sensitivity to infant cues.
Time Frame: 2-hour period
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: dyads
Groups:
- Breast- Versus Bottle-feeding Conditions: This was a within-subject study; all infants were exposed to both conditions: breastfeeding versus bottle-feeding with expressed breast milk
  Order of presentation was counterbalanced.
Arm/Group | Breast- Versus Bottle-feeding Conditions
Number analyzed (Participants) | 94
Number analyzed (dyads) | 47
units on a scale
  Breastfeeding Condition | 14.7 (0.2)
  Bottle-feeding Condition | 14.3 (0.2)
Statistical Analysis 1: Comparison: Breast- Versus Bottle-feeding Conditions; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.115, Mixed Models Analysis; All models adjusted for order of conditions, time since last feeding and infant age

ADVERSE EVENTS:
Time Frame: For the duration of each participant's participation in the study: ~1 week
Description: Definition of adverse event and/or serious adverse event does not differ from the clinicaltrials.gov definitions.
Groups:
- Breastfeeding Condition - Mothers; Breastfeeding Condition - Infants: Mother-infant dyads were observed while breastfeeding during one visit to our laboratory and bottle-feeding expressed breast milk during the other. All mother-infant dyads participated in both conditions. Adverse Event data are reported for mothers (n = 47) and infants (n = 47) separately.
- Bottle-feeding Condition - Mothers; Bottle-feeding Condition - Infants: Mother-infant dyads were observed while bottle-feeding expressed breast milk during one visit to our laboratory and breastfeeding during the other. All mother-infant dyads participated in both conditions. Adverse Event data are reported for mothers (n = 47) and infants (n = 47) separately.
Arm/Group | Breastfeeding Condition - Mothers | Breastfeeding Condition - Infants | Bottle-feeding Condition - Mothers | Bottle-feeding Condition - Infants
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47 | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47 | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/47 | 0/47 | 0/47 | 0/47

LIMITATIONS AND CAVEATS:
This study consisted of mothers who were exclusively or predominantly breastfeeding and who fed expressed breast milk (not formula) when bottle-feeding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT03704051/Prot_SAP_ICF_000.pdf